CLINICAL TRIAL: NCT06470282
Title: Phase Ib/II Study of Enfortumab Vedotin and Pembrolizumab Combined With Radiotherapy as a Bladder-Sparing Trimodality Therapy in Muscle Invasive Bladder Cancer
Brief Title: Enfortumab Vedotin and Pembrolizumab Combined With Radiotherapy in Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Astellas Pharma Inc (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Vadim S Koshkin, Principal Investigator, IND Holder, University of California, San Francisco
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24522; NCI-2024-04701 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer; Muscle-Invasive Bladder Carcinoma; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — enfortumab vedotin; pembrolizumab; Radiotherapy, Intensity-Modulated; Transurethral Resection of Bladder; Cystoscopy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Level 1: 0.75 mg/kg Enfortumab Vedotin (Starting Dose) (Experimental): Participants receive 0.75 mg/kg enfortumab vedotin intravenously (IV) over 30 minutes on days 1 and 8 of cycles 1-5 and pembrolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 5 cycles of enfortumab vedotin and up to 17 cycles of pembrolizumab in the absence of disease progression or unacceptable toxicity. Beginning on cycle 1 day 1, participants also undergo standard of care intensity modulated radiation therapy (IMRT) once daily (QD) for 32 days over 6.5-8 weeks. Participants also undergo TURBT, cystoscopy, as well as imaging throughout the study.
  Interventions: Drug: Enfortumab Vedotin; Biological: Pembrolizumab; Radiation: Intensity Modulated Radiation Therapy (IMRT); Procedure: Transurethral Resection of Bladder Tumor; Procedure: Cystoscopy (CS); Procedure: Computed Tomography (CT); Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET)
- Dose Level 2: 1.0 mg/kg Enfortumab Vedotin (Experimental): Participants receive 1.05 mg/kg enfortumab vedotin intravenously (IV) over 30 minutes on days 1 and 8 of cycles 1-5 and pembrolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 5 cycles of enfortumab vedotin and up to 17 cycles of pembrolizumab in the absence of disease progression or unacceptable toxicity. Beginning on cycle 1 day 1, participants also undergo standard of care intensity modulated radiation therapy (IMRT) once daily (QD) for 32 days over 6.5-8 weeks. Participants also undergo TURBT, cystoscopy, as well as imaging throughout the study.
  Interventions: Drug: Enfortumab Vedotin; Biological: Pembrolizumab; Radiation: Intensity Modulated Radiation Therapy (IMRT); Procedure: Transurethral Resection of Bladder Tumor; Procedure: Cystoscopy (CS); Procedure: Computed Tomography (CT); Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET)
- Dose Level 3: 1.25 mg/kg Enfortumab Vedotin (Experimental): Participants receive 1.25 mg/kg enfortumab vedotin intravenously (IV) over 30 minutes on days 1 and 8 of cycles 1-5 and pembrolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 5 cycles of enfortumab vedotin and up to 17 cycles of pembrolizumab in the absence of disease progression or unacceptable toxicity. Beginning on cycle 1 day 1, participants also undergo standard of care intensity modulated radiation therapy (IMRT) once daily (QD) for 32 days over 6.5-8 weeks. Participants also undergo TURBT, cystoscopy, as well as imaging throughout the study.
  Interventions: Drug: Enfortumab Vedotin; Biological: Pembrolizumab; Radiation: Intensity Modulated Radiation Therapy (IMRT); Procedure: Transurethral Resection of Bladder Tumor; Procedure: Cystoscopy (CS); Procedure: Computed Tomography (CT); Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET)
- Dose Expansion; Recommended Phase 2 Dose (RP2D) (Experimental): Participants receive RP2D of enfortumab vedotin intravenously (IV) over 30 minutes on days 1 and 8 of cycles 1-5 and pembrolizumab IV on day 1 of each cycle. Cycles repeat every 21 days for up to 5 cycles of enfortumab vedotin and up to 17 cycles of pembrolizumab in the absence of disease progression or unacceptable toxicity. Beginning on cycle 1 day 1, participants also undergo standard of care intensity modulated radiation therapy (IMRT) once daily (QD) for 32 days over 6.5-8 weeks. Participants also undergo TURBT, cystoscopy, as well as imaging throughout the study.
  Interventions: Drug: Enfortumab Vedotin; Biological: Pembrolizumab; Radiation: Intensity Modulated Radiation Therapy (IMRT); Procedure: Transurethral Resection of Bladder Tumor; Procedure: Cystoscopy (CS); Procedure: Computed Tomography (CT); Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Enfortumab Vedotin — Given intravenously (IV)
  Other Names: Padcev
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda
Radiation: Intensity Modulated Radiation Therapy (IMRT) — Undergo standard of care, IMRT
  Other Names: Standard of care IMRT
Procedure: Transurethral Resection of Bladder Tumor — Undergo TURBT
  Other Names: Transurethral resection (TURBT)
Procedure: Cystoscopy (CS) — Undergo cystoscopy
  Other Names: CS
Procedure: Computed Tomography (CT) — Undergo CT imaging
  Other Names: CT Scan
Procedure: Magnetic Resonance Imaging (MRI) — Undergo MRI imaging
  Other Names: MRI Scan
Procedure: Positron Emission Tomography (PET) — Undergo PET Scan, may be combined with CT (PET/CT)
  Other Names: PET Scan

SUMMARY:
This phase Ib/II trial studies the side effects, best dose, and effectiveness of enfortumab vedotin (EV) in combination with pembrolizumab and radiation therapy for treating patients with muscle invasive bladder cancer. Standard of care treatment for muscle invasive bladder cancer is chemotherapy, to shrink the tumor before the main treatment is given (neoadjuvant), followed by surgery to remove all of the bladder as well as nearby tissues and organs (radical cystectomy). In cases where patients are not candidates for the standard of care approach or prefer a bladder sparing option, tri-modality therapy with transurethral resection of bladder tumor (TURBT) followed by combined chemotherapy and radiation therapy is used. Enfortumab vedotin is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of tumor cells. Enfortumab attaches to a protein called nectin-4 on tumor cells in a targeted way and delivers vedotin to kill them. It is a type of antibody-drug conjugate. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Intensity-modulated radiation therapy is a type of 3-dimensional radiation therapy that uses computer-generated images to show the size and shape of the tumor. Thin beams of radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor. Giving enfortumab vedotin with pembrolizumab and radiation therapy may work better in treating patients with muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) of enfortumab vedotin given in combination with pembrolizumab and concurrent radiation therapy (RT). (Phase Ib).

II. To assess the toxicity and safety of enfortumab vedotin given in combination with pembrolizumab and concurrent radiation therapy (RT). (Phase Ib).

III. To evaluate the rate of clinical complete response to treatment (cCR) at the RP2D based on 6-month post-treatment cystoscopy, TURBT, cytology, and cross sectional imaging. (Phase II).

IV. To characterize the safety of enfortumab vedotin at the RP2D given in combination with pembrolizumab and concurrent radiation therapy (RT). (Phase II).

SECONDARY OBJECTIVES:

I. To evaluate the rate of cCR 6 months post-treatment start based on cystoscopy, TURBT, and cross sectional imaging. (Phase Ib) II. To evaluate the preliminary efficacy of enfortumab vedotin given in combination with pembrolizumab and concurrent radiation therapy (RT) as measured by 1-year recurrence free survival rate, 2-year cystectomy-free survival rate, 2-year overall survival rate, the median recurrence free survival (RFS) rate, median overall survival, and median cystectomy-free survival. (Phase Ib and Phase II) III. To assess the downstaging to ≤ pT1N0 pT1 or less following completion of treatment, based on 6-month post-treatment cystoscopy, for participants treated at RP2D of enfortumab vedotin (EV). (Phase Ib and Phase II) IV. To assess the downstaging to ≤ pT1N0 or less following completion of treatment, based on 6-month post-treatment cystoscopy, for participants across all EV dose levels. (Phase Ib and Phase II).

EXPLORATORY OBJECTIVES:

I. Assessment of change in tumor gene expression signatures using single-cell ribonucleic acid (RNA) sequencing (scRNA-Seq) following initiation of combination treatment.

II. Assessment of the change in the populations of tumor-infiltrating immune cells (TIICs) induced by initiation of the combination treatment.

III. Determination of the impact of EV/pembrolizumab combination treatment on programmed death-ligand 1 (PD-L1) expression in tumor cells and TIICs, as well as on other immunologic predictive markers.

IV. Assessment of modulation of tumor microenvironment pre- and post-initiation of combination treatment using multiplex immunohistochemistry (IHC).

V. Assessment of the modulation of circulating immune cells following initiation of combination treatment using mass cytometry (cytometry by time of flight, or CyTOF).

VI. Assessment of the change in T-cell receptor repertoire by scRNA-Seq following initiation of combination treatment.

VII. Change in tumor expression of nectin cell adhesion molecule 4 (Nectin-4) following combination treatment relative to baseline.

VIII. Assessment in the change in CD3+ T cell density (T cell count/μm^2) from baseline biopsy to post-RT biopsy in participants with residual tumor, across all EV dose levels and at RP2D.

OUTLINE:

This is a phase Ib, dose escalation study of enfortumab vedotin followed by a phase II study.

Participants receive enfortumab vedotin and pembrolizumab for up to 5 cycle of enfortumab vedotin and up to 17 cycles of pembrolizumab in the absence of disease progression or unacceptable toxicity. Beginning on cycle 1 day 1, participants also undergo non-investigational, standard of care intensity modulated radiation therapy (IMRT) over 6.5-8 weeks.

After completion of study treatment, participants are followed up at 90 days and then every 12 weeks for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed muscle-invasive bladder cancer (cT2,T3,T4a). (Note: Tissue samples are required.) (Participants with cT3/T4a staged disease will be capped at 25% of patients treated at RP2D).
* Urothelial-predominant histology. Mixed histologies other than small cell/neuroendocrine are allowed as long as some urothelial histology is present. Neuroendocrine histology of any component and pure variant (non-urothelial) histology tumors will be excluded. (Patients with < 50% urothelial histology will be capped at 25% of patients treated at RP2D).
* Must be judged by the investigator to be ineligible for radical cystectomy or electing not to undergo radical cystectomy.
* Must be eligible for and agree to receive bladder irradiation as determined by the treating investigator.
* Must have a TURBT within 8 weeks of combination treatment start with viable tumor content. If no viable tumor content is present on TURBT, the patient will be replaced in the study.
* Patients who have autoimmune disease will be evaluated on a case-by-case basis and can only enroll so long as participants are not on active immunosuppression with a corticoid steroid allowance exceeding 10mg of prednisone or equivalent per day.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1.
* Absolute neutrophil count ≥ 1,500/microliter (mcL).
* Platelets >= 100,000/mcL.
* Hemoglobin >= 9.0 g/dL or ≥ 5.6 mmol/L.

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Total bilirubin <= 1.5 × upper limit of normal, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) <= 2.5 X institutional upper limit of normal.
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT)) <= 2.5 X institutional upper limit of normal.
* Creatinine clearance glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2, calculated by Cockcroft-Gault or measured using 24-hour creatinine clearance.
* International normalized ratio (INR) OR prothrombin time (PT) <= 1.5 × upper limit of normal (ULN).

  * If participant is receiving anticoagulant therapy, as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants, participant is eligible.
* Activated partial thromboplastin time (aPTT) <= 1.5 × ULN.

  * If participant is receiving anticoagulant therapy, as long as PT or aPTT is within therapeutic range of intended use of anticoagulants, participant is eligible.
* Ability to understand and the willingness to sign a written informed consent document.
* Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Participants who are hepatitis B virus surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) anti-viral therapy for at least 4-weeks, and have undetectable HBV viral load prior to randomization. Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

  * Note: Hepatitis B screening tests are not required unless patients have a known history of HBV infection.
* Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.

  * Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to cycle 1 day 1.
* Women of child-bearing potential and men with sexual partners of childbearing potential must agree to use adequate contraception for the duration of study participation. Enfortumab vedotin (EV) may cause fetal harm. Women of child-bearing potential must use contraception during treatment with EV and for 120 days after the last dose. Men with female partners who are women of child-bearing potential must use contraception during treatment with EV and for 120 days after the last dose. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Acceptable methods include barrier method, hormonal method, as well as intrauterine devices
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 8 weeks after last administration of study treatment.

Exclusion Criteria:

* Presence of distant metastases on imaging (M1 disease).
* Presence of lymph nodes concerning for regional disease spread (lymph node (LN) > 1.0 cm on short axis present on cross sectional imaging) that is attributable to cancer spread (≥ N1 disease).
* Presence of small cell / neuroendocrine histology in tumor sample (any content).
* Absence of urothelial histology in TURBT tumor sample (pure variant histology).
* Presence of untreated upper tract urothelial cancer.
* Presence of moderate/severe hydronephrosis.
* Presence of extensive carcinoma in situ (CIS).
* Baseline neuropathy grade 2 (G2) or greater.
* Baseline uncontrolled diabetes mellitus.Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥ 8% or HbA1c 7 to < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.

  * Note: Patients with prior diagnosis but with disease under control are eligible
* Prior treatment with systemic immunotherapy or chemotherapy for urothelial cancer.* Note: Prior bacillus calmette-guerin (BCG) and intravesical treatments are allowed
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to cycle 1 day 1.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has received prior radiotherapy within 2 weeks of cycle 1 day 1 or radiation-related toxicities requiring corticosteroids.

  * Note: Two weeks or fewer of palliative radiotherapy for non-central nervous system (CNS) disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention.

  * Note: Administration of killed vaccines is allowed. Any licensed coronavirus 2019 (COVID-19) vaccine (including for emergency use) is allowed in the study as long as they are messenger ribonucleic acid (mRNA) vaccines, replication-incompetent adenoviral vaccines, or inactivated vaccines.
* Major surgery within 2 weeks prior to first dose of EV.

  * Note: Cataract surgery, standard tissue biopsies, and standard of care cardiac devices, such as a pacemaker or stent placed on an elective basis, are allowable procedures.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

  * Note: Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤ 6, and prostate specific antigen (PSA) < 10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis.

  * Note: Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* History of another significant life-limiting malignancy within 2 years prior to the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy.

  * Note: Patients with nonmelanoma skin cancer, curatively treated localized prostate cancer, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Hypersensitivity to pembrolizumab or enfortumab vedotin, or any of their excipients.
* Prior allogeneic stem cell or solid organ transplant.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* History of hepatitis B with detectable HBV viral load (participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization) or known active hepatitis C virus (defined as detectable HCV RNA .[qualitative]) infection.

  * Note: Testing for hepatitis B or C is not required unless clinically indicated or if there is a known history of hepatitis infection
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has had an allogenic tissue/solid organ transplant.
* Pregnant and chest feeding participants are excluded from this study because targeted chemotherapy and radiation have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EV+pembrolizumab, breastfeeding should be discontinued if the mother is treated with these investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) (Phase Ib) | Up to 72 days
  The RP2D is the last dose cohort at which no more than one instance of a dose limiting toxicity (DLT) is observed among 6 participants treated. If the maximum tolerated dose (MTD) cannot be determined due to lack of DLT during the DLT window, the maximum dose level of enfortumab vedotin administered during the study will be declared the RP2D. For the purposes of this study, the RP2D is the MTD.
Proportion of participants reporting dose limiting toxicities (DLTs) (Phase Ib) | Up to 72 days
  The DLT evaluation period will be within the first three cycles (e.g., 56 days or eight weeks, and not to exceed 72 days) of treatment start with enfortumab-vedotin, pembrolizumab, and standard of care fractionation radiation therapy. Participants who receive > 75% of intended enfortumab vedotin, pembrolizumab, and standard of care radiation doses will be considered DLT evaluable (DE).
Frequency of treatment-emergent adverse events | Up to 14 months
  The frequency of adverse events by highest grade and overall attribution to study drugs, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Percentage of participants with Clinical complete response (cCR) (Phase II) | Up to 6 months
  The rate of clinical complete response to treatment (cCR) will be measured as the percentage of participants with cCR based on cystoscopy and TURBT done at 6 months from treatment start. cCR is defined as no visual tumor AND no histological presence of tumor (i.e., ypT0).

SECONDARY OUTCOMES:
Proportion of participants with Clinical Complete Response (cCR) (Phase Ib) | Up to 6 months
  cCR is defined as no visual tumor AND no histological presence of tumor (i.e., ypT0). The point estimate of the clinical complete response (CR) rate will be obtained with 95% confidence interval by Wilson Score confidence interval method
Median Recurrence Free Survival Rate (RFS) at 1 year | Up to 1 year
  The median 1-year RFS is defined as the time of treatment start until evidence of disease recurrence, time of death, or until the participants completes study follow up participation, or is documented as lost to follow up per institutional standard (whichever is sooner) at 1 year determined by Kaplan Meier method.
Median Cystectomy Free Survival rate (CFS) at 2 years | Up to 2 years
  The median 2-year CFS is defined as the time of treatment start until time of cystectomy, time of death, or until the participant completes study follow up participation, or is documented as lost to follow up per institutional standard (whichever is sooner) at 2 years determined by Kaplan Meier method.
Median Overall Survival (OS) at 2 years | Up to 2 years
  The median 2-year OS is defined as the time from start of treatment, across all EV dose levels and at RP2D until time of death, or until the participant is documented as lost to follow up per institutional standard at 2 years determined by Kaplan Meier method.
Median Overall OS | Up to 5 years
  The median overall OS is defined as the time from treatment start until evidence of disease recurrence, time of death, or until the participant completes study follow up participation, or is documented as lost to follow up per institutional standard (whichever is sooner) will be reported.
Median Overall RFS | Up to 5 years
  The median overall RFS is defined as the time from treatment start until evidence of disease recurrence, time of death, or until the participant completes study follow up participation, or is documented as lost to follow up per institutional standard (whichever is sooner) will be reported.
Median Overall CFS | Up to 5 years
  The median overall CFS is defined as the time from treatment start until time of cystectomy, time of death, or until the participant completes study follow up participation, or is documented as lost to follow up per institutional standard (whichever is sooner) will be reported
Proportion of participants who have been downstaged to <= pT1N0, pT1 or less | Up to 6 months
  The point estimate of the proportion of the participants with downstaging to <= pT1N0, pT1, or less at 6 months following the start of treatment will be obtained with 95% confidence interval by Wilson Score confidence interval method.
Proportion of participants who have been downstaged to <= pT1N0 | Up to 6 months
  The point estimate of the proportion of the participants with downstaging to <= pT1N0 at 6 months following the start of treatment will be obtained with 95% confidence interval by Wilson Score confidence interval method.

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Koshkin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No